CLINICAL TRIAL: NCT01223521
Title: Systematic Provision of Intrauterine Contraception After First Trimester Abortion - Effects on Quality of Life and Risk of Repeat Abortion. A Randomized, Prospective Trial.
Brief Title: Intrauterine Contraception After First Trimester Abortion - Effects on Quality of Life and Risk of Repeat Abortion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: City of Helsinki (Other)
Responsible Party: Principal Investigator, Elina Pohjoranta, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TYH2010224
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Contraception
Keywords: Contraception; Abortion; First trimester; Intrauterine device

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate intrauterine contraception (Experimental): IUD (either Cu-IUD or LNG-IUS) inserted immediately after abortion.
  Interventions: Device: Immediate intrauterine contraception
- Control group (No Intervention): Post-abortal contraception is prescribed by the hospital but on the responsibility of the patient.

INTERVENTIONS:
Device: Immediate intrauterine contraception — A Cu-IUD or LNG-IUS is inserted after abortion.
  Arms: Immediate intrauterine contraception

SUMMARY:
A randomized prospective study on the effects of immediate provision of intrauterine contraception after first trimester induced abortion - effects on repeat abortions and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Duration of pregnancy < 12 weeks.
* Age ≥18 years

Exclusion Criteria:

* Contraindication for spiral insertion: uterine anomaly, infection, copper allergy (Cu-IUD).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2010-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of repeat abortions | 5 years
  Number of subsequent abortions during five years follow-up time.

CONTACTS AND LOCATIONS:
Overall Officials: Oskari Heikinheimo, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Satu P Suhonen, MD, PhD, Study Director — City of Helsinki
Locations (1):
- Dept Obstetrics and Gynecology, Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pohjoranta E, Mentula M, Gissler M, Suhonen S, Heikinheimo O. Provision of intrauterine contraception in association with first trimester induced abortion reduces the need of repeat abortion: first-year results of a randomized controlled trial. Hum Reprod. 2015 Nov;30(11):2539-46. doi: 10.1093/humrep/dev233. Epub 2015 Sep 14. PMID 26370664
- [Background] Toffol E, Pohjoranta E, Suhonen S, Hurskainen R, Partonen T, Mentula M, Heikinheimo O. Anxiety and quality of life after first-trimester termination of pregnancy: a prospective study. Acta Obstet Gynecol Scand. 2016 Oct;95(10):1171-80. doi: 10.1111/aogs.12959. PMID 27500660
- [Background] Pohjoranta E, Suhonen S, Mentula M, Heikinheimo O. Intrauterine contraception after medical abortion: factors affecting success of early insertion. Contraception. 2017 Mar;95(3):257-262. doi: 10.1016/j.contraception.2016.10.012. Epub 2016 Nov 9. PMID 27836586
- [Derived] Pohjoranta E, Suhonen S, Gissler M, Ikonen P, Mentula M, Heikinheimo O. Early provision of intrauterine contraception as part of abortion care-5-year results of a randomised controlled trial. Hum Reprod. 2020 Apr 28;35(4):796-804. doi: 10.1093/humrep/deaa031. PMID 32266392
- [Derived] Pohjoranta E, Mentula M, Suhonen SP, Heikinheimo O. Predicting poor compliance with follow-up and intrauterine contraception services after medical termination of pregnancy. BMJ Sex Reprod Health. 2018 Sep 15:bmjsrh-2018-200098. doi: 10.1136/bmjsrh-2018-200098. Online ahead of print. PMID 30219793